CLINICAL TRIAL: NCT05904756
Title: Patient Satisfaction and Oral Healthy Related Quality of Life of Polyetherketoneketone and Metal Framework for All-on-four Implant Supported Fixed Detachable Prosthesis: A Crossover Study.
Brief Title: Patient Satisfaction and Oral Healthy Related Quality of Life of Polyetherketoneketone and Metal Framework.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Elsawy, lecturer, Department of prosthodontics, principle investigator, Mansoura University
Other Study IDs: A0105023RP
Record Dates: First submitted 2023-06-06; First posted 2023-06-15 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Metal framework group: Two sets of patients were made (10 patients/set) using random-generated numbers created by a computer program (Excel sheet). Conventional complete denture will be fabricated first and patient will wear the denture for 3 months. Then 4 implants will be placed according to all in 4 concept.after 3 months of asseointegration,the first 10 participants will recieve metal framework first. After 3 months, patient satisfaction and oral healthy related quality of lifewill be measured.
  Interventions: Device: framework for implant supported prosthesis, fabricated from metal of polyetherketoneketone
- PEKK framework group: metal framework will be replaced by PEKK framework. After another 3 months, measurements will be repeated. The second 10 patients received polyetherketoneketone first, and after 3 months, measurements will be made. Then, polyetherketoneketone framework will be replaced by Metal framework and measurements( Patient satisfaction and oral healty related quality of life) will be repeated after another 3 months in across over design.
  Interventions: Device: framework for implant supported prosthesis, fabricated from metal of polyetherketoneketone

INTERVENTIONS:
Device: framework for implant supported prosthesis, fabricated from metal of polyetherketoneketone — evaluation of patient satisfaction and oral healty related quality of life

SUMMARY:
The patients' satisfaction and oral health related quality of life (OHRQL) of different framework material remains uncertain. Thus, the aim of this clinical cross over study was to compare patient satisfaction and OHRQL OF polyetherketoneketone and metal framework for All-on-four implant supported fixed prosthesis

DETAILED DESCRIPTION:
10 completely edentulous patients around age of 50-60 years will be selected for this study from the Outpatient Clinic, Faculty of Dentistry, Mansoura University.

All selected participants will receive a new complete dentures (CD) fabricated with bilateral balanced occlusion utilizing semi-anatomical acrylic teeth. The patients were instructed to wear the dentures for 3 months to develop adequate neuromuscular control, and then, clinical performance and patient satisfaction will be evaluated.

Each participant will receive 4 implants according to the "All-on-4 concept," and the implants will be immediately loaded with mandibular denture. Three months after osseointegration, patients received a definitive fixed detachable prosthesis either from PEKK or metal with composite teeth in a crossover designs. Two sets of patients will be made (10 patients/set) using random-generated numbers created by a computer program (Excel sheet). The first 10 participants will recieve metal framework first. After 3 months, patient satisfaction and OHRQoL will be measured and metal framework will be replaced by PEKK framework. After another 3 months, measurements will be repeated. The second 10 patients received PEKK first, and after 3 months, measurements will be made. Then, PEKK framework was replaced by Metal framework and measurements were repeated after another 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient available restorative space (from the proposed occlusal plane to soft tissue • covering residual ridge) of at least 20 mm to accommodate all types of tested prosthesis.
* They had completely edentulous maxilla and mandible at least six months after the last extraction.
* Sufficient residual alveolar ridge quantity and quality (D2-D3)
* Maxillary and mandibular residual alveolar ridges covered by healthy non-inflamed mucosa with even compressibility.
* Normal maxillo-mandibular relationship.

Exclusion Criteria:

All diseases or syndromes are contraindicated with implant surgery such as:

* General contraindications for surgical procedures such as patients with head and neck radio therapy, patients with bleeding disorders, hepatic patients.
* Patients with metabolic disorders that affect Osseo integration such as diabetes mellitus, and osteoporosis.
* Long term immunosuppressive and corticosteroid drug therapy.
* Abnormal detrimental habits, e.g. bruxism and clenching.
* Heavy smokers and alcoholic patients.
* All patients will be informed about the steps involved in this research and they will sign a

written consent form of the ethical committee of faculty of dentistry Mansoura University for approval to take part in this research and come to the follow up visits.

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Sample size calculation was based on difference in OHIP between CD & MB groups retrived from previous research using 2-tailed test , α error =0.05 and power = 90.0% , the total calculated sample size will be 10 cases in each group.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-01-04 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
The patients' satisfaction using a visual analog scale (VAS) | 1 year
  VAS score include, comfort with prosthesis, ease of cleaning appearance, decreased embarrassment, ease of speaking, general satisfaction of mandibular prosthesis compared to teeth and prosthesis apart of you, and decreased embracing. Higher score indicating increase satisfaction, and lower scores indicating less satisfaction.

SECONDARY OUTCOMES:
Oral healthy related quality of life (OHRQoL) | 1 year
  The arabic version of OHRQoL such as, functional limitation, physical pain, psychologic discomfort, psychologic disability, and social disability. For each item of the 14 items were never (= 1), hardly ever (= 2), occasionally (= 3), fairly often (= 4), and very often (= 5). Lower scores indicated higher OHRQoL, vice versa

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed E Sawy, Study Director — Mansoura University
Locations (1):
- Faculty of dentistry , Mansoura University, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No